CLINICAL TRIAL: NCT02592174
Title: Prevalence, Characteristics and Risk Factors of HIV-Associated Neurocognitive Disorders in Subjects Between the Ages of 55 and 70 Years: An Exposed/Unexposed Cross Sectional Study
Acronym: HAND55-70
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS EP58 HAND 55-70
Record Dates: First submitted 2015-10-20; First posted 2015-10-30 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Quality of Life; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV subjects (Other): * Evaluation of health-related quality of life and collection of social and demographic informations at the inclusion visit.
  * Neurocognitive assessment with neuropsychologist and walking speed, grasp force and one leg stand assessments at the neurocognitive visit.
  * Two substudies will be proposed:
    * cerebral images sub-study (80 patients in the centers of Montpellier and the centers of Nîmes)
    * sub-study on immune activating markers with sample's collection (plasma), 85 patients in the centers of Montpellier and the centers of Nîmes.
  Interventions: Other: Health related quality of life and social and demographic informations; Other: Neurocognitive assessment; Radiation: cerebral images sub-study

INTERVENTIONS:
Other: Health related quality of life and social and demographic informations — At the inclusion visit with a self-assessment questionnaire
Other: Neurocognitive assessment — At the neurocognitive visit, with standard test as CONSTANCES cohort
Radiation: cerebral images sub-study — Standard magnetic resonance imaging

SUMMARY:
The primary objective is to measure the prevalence of according to the Frascati classification in a HIV-infected population aged between 55 and 70 years (exposed group) and to compare it with the prevalence of HIV-Associated Neurocognitive Disorders (HAND) in unexposed subjects from the general population-based cohort CONSTANCES, matching subjects on age, gender, geographical origin and socioprofessional category.

DETAILED DESCRIPTION:
Secondary objectives are:

* To study factors associated with Asymptomatic Neurocognitive Impairment (ANI) or Mild Neurocognitive Disorders (MND) by distinguishing the impact of traditional risk factors of neurocognitive impairment and those related to HIV infection,
* To compare in the exposed and unexposed population physical characteristics, complaints and comorbidities,
* To compare global neurocognitive scores in both populations after standardized normal reduction of each test.

Methodology:

HIV-infected subjects aged between 55 and 70 years will be recruited in centres that support people who living with HIV usually. The study will be proposed consecutively to all subjects aged between 55 and 70 year. A brief inquiry will collect motives on subjects that refuse to participate. A minimum of 70 subjects by 5 years age categories will be included. Unexposed subjects will be recruited in the same regions as their HIV-infected counterparts from the CONSTANCES database, a general population health cohort, after random selection matched on age, gender, geographical origin and socioprofessional category (2 HIV-unexposed subjects for 1 exposed subject). Data collection will follow the same methods as in the CONSTANCES cohort, in particular the neurocognitive tests by trained neuropsychologists.

ELIGIBILITY:
For the HIV-infected, inclusion criteria are:

* An age between 55 and 70 years including,
* A HIV-viral load <50 copies/mL for at least 24 months (with a minimum of three viral loads during the 24 months period, and a last viral load within 6 months of inclusion). Blips, defined by a transitory elevation of viral load < 200 copies/ml, are not considered as an exclusion criteria if objectified twice or less during the 24 months period,
* A CD4 cells level ≥ 200 cells/µL during the 12 months preceding inclusion, with a last CD4 cells value < 6 months from inclusion,
* free and informed consent,
* Patient enrolled in or a beneficiary of a Social Security programme (State Medical Aid is not a Social Security programme)

Non-inclusion criteria are:

* Delirium or active central nervous system disease
* Major psychiatric disease, sensory loss, illiteracy, language barrier inducing difficulties in neurocognitive assessment,
* Neurocognitive extensive evaluation in the last 6 months,
* History of neurological disease with clinical sequels,
* Subjects participating in a study excluding participating in another study,
* Vulnerability, such as an age under 18, tutorship, guardianship, or subjects deprived of liberty by a legal or administrative decision.

Inclusion criteria for the subjects from the CONSTANCES cohort are an age between 55 and 70 years. Non-inclusion criteria are the same as the HIV-infected subjects, as well as reported HIV-infection or antiretroviral treatment.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
The Prevalence of Neurocognitive troubles HAND in the HIV-infected and to compare it with the prevalence in the HIV-unexposed population in the CONSTANCES cohort. | at month 3 (neurocognitive evaluation)
  Neurocognitive assessment with neuropsychologist and walking speed, grasp force and one leg stand assessments at month 3 (the neurocognitive visit).

SECONDARY OUTCOMES:
The prevalence of Asymptomatic Neurocognitive Impairment (ANI) | at month 3 (neurocognitive evaluation)
  Neurocognitive assessment with neuropsychologist and walking speed, grasp force and one leg stand assessments at month 3 (the neurocognitive visit).
The prevalence of HIV-Associated Dementia(HAD) | at month 3 (neurocognitive evaluation)
  Neurocognitive assessment with neuropsychologist and walking speed, grasp force and one leg stand assessments at month 3 (the neurocognitive visit).
The prevalence of Mild Neurocognitive Disorder (MND) | at month 3 (neurocognitive evaluation)
  Neurocognitive assessment with neuropsychologist and walking speed, grasp force and one leg stand assessments at month 3 (the neurocognitive visit).
Cognitive score distributions untreated or after transformation according to their distribution characteristics | at month 3 (neurocognitive evaluation)
Physical score distributions untreated or after transformation according to their distribution characteristics | at month 3 (neurocognitive evaluation)
A comparison of a global cognitive score in both populations after standardized normal reduction of each test. | at month 3 (neurocognitive evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Berr, Study Director — Inserm U1061
Locations (6):
- France (6):
  - Centre Hospitalier de Cannes - Service de Médecine Interne Oncologie, Cannes
  - Hôpital Michallon- Service des Maladies Infectieuses, Grenoble
  - Hôpial Sainte Marguerite - Service d'hématologie-Cisih, Marseille
  - Hôpital Gui de Chauliac - Service des Maladies Infectieuses, Montpellier
  - Hôpital Carémeau - Service des Maladies Infectieuses, Nîmes
  - Hôpital Bretonneau - Service des Maladies Infectieuses, Tours

REFERENCES:
- [Derived] Makinson A, Dubois J, Eymard-Duvernay S, Leclercq P, Zaegel-Faucher O, Bernard L, Vassallo M, Barbuat C, Geny C, Thouvenot E, Costagliola D, Ozguler A, Zins M, Simony M, Reynes J, Berr C. Increased Prevalence of Neurocognitive Impairment in Aging People Living With Human Immunodeficiency Virus: The ANRS EP58 HAND 55-70 Study. Clin Infect Dis. 2020 Jun 10;70(12):2641-2648. doi: 10.1093/cid/ciz670. PMID 31755936